CLINICAL TRIAL: NCT01416584
Title: A Bridge to Treatment: The Therapeutic Workplace and Methadone Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00020746; R01DA023864 (NIH)
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Opiate Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care Control (No Intervention): Participants in this group were offered employment in the Therapeutic Workplace without urinalysis testing or the methadone treatment requirement. They were offered the methadone treatment but were not required to join in order to gain access to the workplace.
- Methadone Contingency Group (Experimental): Participants in this group were allowed to work and earn wages as long as they enrolled in the methadone treatment and continued to take does of methadone consistently (employment-based reinforcement).
  Interventions: Behavioral: methadone contingency
- Methadone & Abstinence Contingency (Experimental): Participants in this group were able to access work if they enrolled in the methadone treatment and consistently took their medication, but they also received a decrease in base pay if they test positive for opiates or cocaine on the drug screens (employment-based reinforcement).
  Interventions: Behavioral: methadone contingency; Behavioral: Methadone & Abstinence Contingency

INTERVENTIONS:
Behavioral: methadone contingency — Participants had to enroll in methadone treatment and take daily doses of methadone to gain access to the workplace.
  Arms: Methadone & Abstinence Contingency; Methadone Contingency Group
Behavioral: Methadone & Abstinence Contingency — Participants had to enroll in methadone treatment and take daily doses of methadone to gain access to the workplace and they had to provide opiate and cocaine negative urine samples to maintain the maximum pay.
  Arms: Methadone & Abstinence Contingency

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the Therapeutic Workplace in promoting methadone treatment and increasing abstinence in unemployed, out-of-treatment injection heroine users.

DETAILED DESCRIPTION:
A randomized study is planned for 5 years to evaluate the effectiveness of the Therapeutic Workplace in promoting methadone treatment and abstinence in unemployed injection drug users. Participants will be recruited through street outreach, at agencies that serve the target populations, and informal word-of-mouth referrals. Participants will be invited to attend the workplace and to enroll in the methadone treatment. To engage participants in the workplace, they will be allowed to work independent of whether they enroll in methadone treatment and independent of their drug use. The workplace participants (N=162) will be randomly assigned to three groups. The "Usual Care Control" participants will be allowed to work independent of their methadone use or urinalysis results. The "Methadone Contingency" participants will be required to take methadone to attend work, and will receive a brief pay decrease for failing to take their medication. The "Methadone & Abstinence Contingency" participants will be required to take their medication in order to attend work, as well as receive a brief pay decrease for any positive urine samples for both cocaine and methadone.

ELIGIBILITY:
Individuals were eligible if they were:

* at least 18 years old,
* reported injection drug use in the past 30 days,
* met the Diagnostic and Statistical Manual (DSM)-IV criteria for opioid dependence,
* reported using heroin at least 21 out of the past 30 days,
* provided an opiate-positive urine sample,
* showed visible signs of injection drug use (i.e., track marks),
* reported not receiving substance abuse treatment in the past 30 days,
* lived in Baltimore,
* and were unemployed.

Participants were excluded if they

* had current severe psychiatric disorders or chronic medical conditions that would interfere with their ability to participate in the workplace,
* reported current suicidal or homicidal ideation,
* had physical limitations that would prevent them from using a keyboard,
* had medical insurance coverage (as this would disqualify them from receiving interim methadone treatment),
* were pregnant or breastfeeding,
* or were currently considered a prisoner.

Eligible participants were invited to participate in a 4-week induction. Participants who attended the workplace for at least five minutes on two out of five workdays in the last week of induction were randomly assigned to one of three conditions and were invited to attend the workplace for an additional 26 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2008-10; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Silverman, Ph.D., Principal Investigator — Professor, Johns Hopkins University School of Medicine
Locations (1):
- Center for Learning and Health, Johns Hopkins Bayview Medical Campus, 5200 Eastern Ave., Suite W142, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holtyn AF, Koffarnus MN, DeFulio A, Sigurdsson SO, Strain EC, Schwartz RP, Leoutsakos JM, Silverman K. The therapeutic workplace to promote treatment engagement and drug abstinence in out-of-treatment injection drug users: a randomized controlled trial. Prev Med. 2014 Nov;68:62-70. doi: 10.1016/j.ypmed.2014.02.021. Epub 2014 Mar 4. PMID 24607365

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through agencies that served the target population, street outreach, and a respondent-driven sampling referral system in which study participants were paid for successfully referring others to the study. Interested individuals completed a brief screening interview that gauged study eligibility.
Pre-assignment Details: Eligible participants were invited to participate in a 4-week induction. During induction, participants were invited to attend the therapeutic workplace. Participants who attended the workplace for at least five minutes on two out of five workdays in the last week of induction were randomly assigned to one of three conditions.
Groups:
- Usual Care Control: Participants in this group were offered employment in the Therapeutic Workplace without urinalysis testing or the methadone treatment requirement. They were offered the methadone treatment but are not required to join in order to gain access to the workplace.
- Methadone Contingency Group: Participants in this group were allowed to work and earn wages as long as they enrolled in the methadone treatment and continued to take does of methadone consistently.
- Methadone & Abstinence Contingency: Participants were be able to access work if they enroll in the methadone treatment and consistently take their medication, but also received a decrease in base pay if they test positive for opiates or cocaine on the drug screens.
Period: Overall Study
Arm/Group | Usual Care Control | Methadone Contingency Group | Methadone & Abstinence Contingency
Started | 30 | 35 | 33
Completed | 27 | 33 | 32
Not Completed | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Usual Care Control: Participants in this group will be offered employment in the Therapeutic Workplace without urinalysis testing or the methadone treatment requirement. They will be offered the methadone treatment but are not required to join in order to gain access to the workplace.
- Methadone Contingency Group: Participants in this group will only be allowed to work and earn wages as long as they enroll in the methadone treatment and continue to take does of methadone consistently.
- Methadone & Abstinence Contingency: Participants will only be able to access work if they enroll in the methadone treatment and consistently take their medication, but also will receive a decrease in base pay if they test positive for opiates or cocaine on the drug screens.
- Total: Total of all reporting groups
Arm/Group | Usual Care Control | Methadone Contingency Group | Methadone & Abstinence Contingency | Total
Number analyzed (Participants) | 30 | 35 | 33 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 34 | 33 | 97
  >=65 years | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (9) | 42 (10) | 44 (9) | 44 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 15 | 33
  Male | 20 | 27 | 18 | 65
Region of Enrollment [Number; unit: participants]
  United States | 30 | 35 | 33 | 98

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Months in Methadone Treatment
Description: The percentage of months in which participants were enrolled in methadone treatment during the 6-month intervention evaluation period?
Time Frame: 6 months
Population: Intent to treat
Measure: Mean (Full Range); unit: percent of months in methadone treatment
Groups:
- Methadone & Abstinence Contingency: Participants in this group were able to access work if they enrolled in the methadone treatment and consistently took their medication, but they also received a decrease in base pay if they test positive for opiates or cocaine on the drug screens.
Arm/Group | Usual Care Control | Methadone Contingency Group | Methadone & Abstinence Contingency
Number analyzed (Participants) | 30 | 35 | 33
percent of months in methadone treatment | 81 [0 to 100] | 82 [0 to 100] | 88 [0 to 100]
Statistical Analysis 1: Comparison: Usual Care Control vs Methadone Contingency Group; Test type: Superiority; p = 0.60, General Estimating Equation (GEE); Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.40 to 4.83]
Statistical Analysis 2: Comparison: Usual Care Control vs Methadone & Abstinence Contingency; Test type: Superiority; p = 0.88, General Estimating Equation (GEE); Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.32 to 3.73]
Statistical Analysis 3: Comparison: Methadone Contingency Group vs Methadone & Abstinence Contingency; Test type: Superiority; p = 0.64, General Estimating Equation (GEE); Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.36 to 4.46]

2. Primary Outcome: Percentage of Monthly Urine Sample Negative for Opiates
Description: Percentage of urine sample negative for opiates at each of the six 30-day assessments scheduled throughout the intervention evaluation
Time Frame: 6 months
Population: Intent to treat
Measure: Mean (Full Range); unit: percentage of opiate negative
Arm/Group | Usual Care Control | Methadone Contingency Group | Methadone & Abstinence Contingency
Number analyzed (Participants) | 30 | 35 | 33
percentage of opiate negative | 54 [0 to 100] | 61 [0 to 100] | 75 [0 to 100]
Statistical Analysis 1: Comparison: Usual Care Control vs Methadone & Abstinence Contingency; Test type: Superiority; p = 0.02, General Estimating Equation (GEE); Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.38 to 0.41]
Statistical Analysis 2: Comparison: Usual Care Control vs Methadone Contingency Group; Test type: Superiority; p = 0.39, General Estimating Equation (GEE); Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.34 to 1.57]
Statistical Analysis 3: Comparison: Methadone Contingency Group vs Methadone & Abstinence Contingency; Test type: Superiority; p = 0.10, General Estimating Equation (GEE); Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.53 to 2.26]

3. Primary Outcome: Percentage of Monthly Urine Samples Negative for Cocaine
Description: Was the participant's urine sample negative for cocaine at each of the six 30-day assessments scheduled throughout the intervention evaluation period?
Time Frame: 6 months
Population: intent to treat
Measure: Mean (Full Range); unit: percentage of cocaine negative
Arm/Group | Usual Care Control | Methadone Contingency Group | Methadone & Abstinence Contingency
Number analyzed (Participants) | 30 | 35 | 33
percentage of cocaine negative | 32 [0 to 100] | 55 [0 to 100] | 57 [0 to 100]
Statistical Analysis 1: Comparison: Usual Care Control vs Methadone & Abstinence Contingency; Test type: Superiority; p = 0.02, General Estimating Equation (GEE); Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.36 to 0.38]
Statistical Analysis 2: Comparison: Usual Care Control vs Methadone Contingency Group; Test type: Superiority; p = 0.02, General Estimating Equation (GEE); Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.38 to 0.41]
Statistical Analysis 3: Comparison: Methadone Contingency Group vs Methadone & Abstinence Contingency; Test type: Superiority; p = 0.85, General Estimating Equation (GEE); Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.20 to 5.66]

4. Secondary Outcome: Percentage of M,W,F Urine Samples Negative for Cocaine
Description: Was each participant's urine sample negative for cocaine at each of the Monday, Wednesday, Friday urine samples scheduled throughout the intervention evaluation period?
Time Frame: 6 months
Population: intent to treat
Measure: Mean (Full Range); unit: percentage of urine samples
Arm/Group | Usual Care Control | Methadone Contingency Group | Methadone & Abstinence Contingency
Number analyzed (Participants) | 30 | 35 | 33
percentage of urine samples | 25 [3.8 to 100] | 44 [0 to 100] | 48 [0 to 100]
Statistical Analysis 1: Comparison: Usual Care Control vs Methadone & Abstinence Contingency; Test type: Superiority; p = 0.01, General Estimating Equation (GEE); Odds Ratio (OR) = 0.35, 95% CI 2-sided [0.34 to 0.35]
Statistical Analysis 2: Comparison: Usual Care Control vs Methadone Contingency Group; Test type: Superiority; p = 0.03, General Estimating Equation (GEE); Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.39 to 0.44]
Statistical Analysis 3: Comparison: Methadone Contingency Group vs Methadone & Abstinence Contingency; Test type: Superiority; p = 0.63, General Estimating Equation (GEE); Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.42 to 1.69]

5. Secondary Outcome: Percentage of M,W,F Urine Samples Negative for Opiates
Description: Was each participant's urine sample negative for opiates at each of the Monday, Wednesday, Friday urine samples scheduled throughout the intervention evaluation period?
Time Frame: 6 months
Population: intent to treat
Measure: Mean (Full Range); unit: percentage of M,W,F urine samples
Arm/Group | Usual Care Control | Methadone Contingency Group | Methadone & Abstinence Contingency
Number analyzed (Participants) | 30 | 35 | 33
percentage of M,W,F urine samples | 43 [3.8 to 100] | 50 [0 to 100] | 65 [0 to 100]
Statistical Analysis 1: Comparison: Usual Care Control vs Methadone & Abstinence Contingency; Test type: Superiority; p = 0.01, General Estimating Equation (GEE); Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.39 to 0.40]
Statistical Analysis 2: Comparison: Usual Care Control vs Methadone Contingency Group; Test type: Superiority or Other; p = 0.37, General Estimating Equation (GEE); Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.36 to 1.55]
Statistical Analysis 3: Comparison: Methadone Contingency Group vs Methadone & Abstinence Contingency; Test type: Superiority; p = 0.05, General Estimating Equation (GEE); Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.28 to 1.00]

6. Other Pre Specified Outcome: Did Participant Share Needles or Works?
Description: Percent of months that participants reported sharing needles or works.
Time Frame: 6 months
Population: Due to the very low rate of reports of sharing needles or works in all groups, we did not analyze this measure. This grant has ended and there is no funding to conduct more analyses.
Arm/Group | Usual Care Control | Methadone Contingency Group | Methadone & Abstinence Contingency
Number analyzed (Participants) | 0 | 0 | 0

7. Other Pre Specified Outcome: Went to Shooting Gallery/House or Other Place Where Users go to Shoot-up?
Description: The percent of months that participants reported going to a shooting gallery/hour or other place where users go to shoot-up.
Time Frame: 6 months
Population: Due to the very low rate of reports of going to a shooting gallery/house or other place where users go to shoot-up in all groups, we did not analyze this measure. This grant has ended and there is no funding to conduct more analyses.
Arm/Group | Usual Care Control | Methadone Contingency Group | Methadone & Abstinence Contingency
Number analyzed (Participants) | 0 | 0 | 0

8. Other Pre Specified Outcome: Did Participant Inject Drugs?
Description: Percent of months that participants reported injecting drugs.
Time Frame: 6 months
Population: We did not analyze this measure. This grant has ended and there is no funding to conduct more analyses.
Arm/Group | Usual Care Control | Methadone Contingency Group | Methadone & Abstinence Contingency
Number analyzed (Participants) | 0 | 0 | 0

9. Other Pre Specified Outcome: In Methadone Treatment at End of Treatment
Description: Was each participant in methadone treatment at the end of the 6-month intervention evaluation period?
Time Frame: 6 months
Population: We did not analyze this measure. This grant has ended and there is no funding to conduct more analyses.
Arm/Group | Usual Care Control | Methadone Contingency Group | Methadone & Abstinence Contingency
Number analyzed (Participants) | 0 | 0 | 0

10. Other Pre Specified Outcome: Entered Methadone Treatment
Description: Did the participant enter methadone treatment at any point in the 6-month treatment period?
Time Frame: 6 months
Population: We did not analyze this measure. This grant has ended and there is no funding to conduct more analyses.
Groups:
- Usual Care Control: Participants could work and earn stipends, but did not have to enter methadone treatment or provide drug-free urine samples to work or earn money.
- Methadone Contingency Group: Participants were required to stay enrolled in methadone treatment to work and earn wages.
- Methadone & Abstinence Contingency: Participants were required to stay enrolled in methadone treatment to work and earn wages and provide urine samples negative for opiates and cocaine to maintain maximum pay.
Arm/Group | Usual Care Control | Methadone Contingency Group | Methadone & Abstinence Contingency
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Usual Care Control | Methadone Contingency Group | Methadone & Abstinence Contingency
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/35 | 1/33
Other Adverse Events (participants affected / at risk) | 0/30 | 1/35 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care Control (N=30) | Methadone Contingency Group (N=35) | Methadone & Abstinence Contingency (N=33)
Hospitalization for car accident (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalization for Vaginal Swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care Control (N=30) | Methadone Contingency Group (N=35) | Methadone & Abstinence Contingency (N=33)
Dizziness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Inpatient heroin detoxification (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No